CLINICAL TRIAL: NCT04678999
Title: Neurobiological Mechanisms of Mind-body Therapy (Remotely Delivered) for Knee Osteoarthritis
Brief Title: Mind-body Therapy (Remotely Delivered) for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13281
Record Dates: First submitted 2020-12-09; First posted 2020-12-22 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Educational Status

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tai Chi (Experimental): The intervention will delivered via a secure Zoom video platform. One of two Tai Chi instructors will teach each of the classes. Tai Chi instructors will be selected prior to study start on the basis of familiarity with our previous Tai Chi protocols and experience working with OA patients.
  Interventions: Behavioral: Mind-body exercise and education
- Wellness Education (Experimental): At each session, a variety of health professionals will provide a didactic lesson on a topic relating to knee OA. An informational brochure on knee OA education is presented to all participants during the first session. Each session will last 60 minutes including a 10-minute instructor-led program of stretching or flexibility exercises via a zoom platform.
  Interventions: Behavioral: Mind-body exercise and education

INTERVENTIONS:
Behavioral: Mind-body exercise and education — The intervention will delivered via a secure Zoom video platform.

SUMMARY:
This proposal aims to provide crucial knowledge about the neurobiological mechanisms underlying Tai Chi mind-body therapy for knee osteoarthritis (OA). The central mechanism of knee OA pain will be investigated using brain imaging technology to evaluate how brain function and structure change in response to mind-body exercise over time.

Sixty eligible individuals who meet the American College of Rheumatology criteria for knee OA will be randomized into Tai Chi or wellness education interventions for 12 weeks. The investigators will compare changes in resting state functional connectivity of the cognitive control network, and functional magnetic resonance imaging responses to pressure pain and brain morphometry, as well as their association with clinical outcomes. The findings will lead to the establishment of a new treatment paradigm in OA and have broad application to the management of chronic musculoskeletal pain.

DETAILED DESCRIPTION:
The study will investigate the central mechanism of knee OA pain using brain imaging technology to evaluate how brain function and structure change in response to mind-body exercise over time. Tai Chi mind body therapy may work by modulating the interaction among cognitive control network, default mode network, descending pain modulation system, limbic system, salient network, and sensory motor system through complex mind-body interactions. By combining multiple brain imaging modalities measurements, investigators will examine the neural substrates of Tai Chi compared with wellness education in adults with knee OA. The investigators will compare changes in resting state functional connectivity of the cognitive control network, brain morphometry and functional magnetic resonance imaging responses to pressure pain, as well as their association with clinical outcomes. Results of this innovative mechanistic study will have important therapeutic implications and provide critical insight into the clinical, behavioral, and neurobiological mechanisms of the potential disease-modifying role of mind-body therapies for knee OA.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years or older
* Unilateral or bilateral Knee OA
* Fulfills the American College of Rheumatology Criteria for symptomatic knee OA
* Willing to undergo MRI at baseline and follow-up
* WOMAC pain subscale score ≥2 on weight-bearing questions

Exclusion Criteria:

* Serious medical conditions limiting ability of patient to participate in the study such as, symptomatic cardiovascular, symptomatic pulmonary disease requiring supplemental oxygen, uncontrolled metabolic diseases, severe renal and liver disease
* Presence of any contraindications to fMRI scanning. Including but not limited to: cardiac pacemaker, metal implants, fear of closed spaces, pregnancy, weight >300 lbs

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
resting state functional connectivity | 12 weeks
  Change in resting state functional connectivity between baseline to 12 weeks as measured by fMRI.

SECONDARY OUTCOMES:
Brain Morphometry | 12 weeks
  Brain morphometry as measured by gray matter volume difference between baseline and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chenchen Wang, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Division of Rheumatology, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No